CLINICAL TRIAL: NCT05070728
Title: A Phase 3, Multicenter, Prospective, Randomized, Masked, Controlled, Safety and Efficacy Study of a Fluocinolone Acetonide (FA) Intravitreal 0.05 mg Insert (Yutiq 0.05 mg) in Subjects With Chronic Non-Infectious Uveitis Affecting the Posterior Segment of the Eye
Brief Title: Safety and Efficacy of an Injectable Fluocinolone Acetonide Intravitreal (FAI) Insert
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No longer pursuing indication
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EYP-2102-001
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Uveitis; Uveitis, Posterior; Uveitis, Intermediate
Keywords: EYP-2102; EyePoint; Uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Posterior; Uveitis, Intermediate | interventions — Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sham Comparator (Sham Comparator): Intravitreal sham injection
  Interventions: Drug: Sham Injector
- FAI insert (0.05 mg fluocinolone acetonide) (Active Comparator): Fluocinolone acetonide (FA) intravitreal 0.05 mg insert (Yutiq 0.05 mg).
  Interventions: Drug: FAI Insert

INTERVENTIONS:
Drug: Sham Injector — Intravitreal sham injection
  Other Names: Sham Comparator
  Arms: Sham Comparator
Drug: FAI Insert — Yutiq 0.05 mg contains 0.05 mg FA and was designed to deliver FA into the vitreous humor for at least 24 weeks.
  Yutiq 0.05 mg was administered to the study eye by injection through the pars plana using a pre-loaded applicator with a 25-gauge needle.
  Other Names: Active Drug
  Arms: FAI insert (0.05 mg fluocinolone acetonide)

SUMMARY:
A study to evaluate the safety and efficacy of a fluocinolone acetonide intravitreal (FAI) insert in the management of subjects with chronic non-infectious uveitis affecting the posterior segment of the eye.

DETAILED DESCRIPTION:
This was a phase 3, multicenter, randomized, masked, controlled study to evaluate the safety and efficacy of an injectable FAI insert for the management of subjects with chronic non-infectious uveitis affecting the posterior segment of the eye. Subjects were randomized to receive either a sham injection or the FAI insert and were observed for 1 year following treatment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or non-pregnant female at least 18 years of age at time of consent.
2. One or both eyes had a history of recurrent non-infectious uveitis affecting the posterior segment of the eye (intermediate, posterior, or panuveitis) with or without anterior uveitis >1 year duration.
3. During the 52 weeks prior to enrollment (Day 1), the subject must have received treatment for uveitis in the study eye with:

   1. Systemic corticosteroid or other systemic therapies for at least 12 consecutive or non-consecutive weeks, AND/OR
   2. at least 2 intra- or peri-ocular administrations of corticosteroid in the study eye, OR
   3. the study eye has experienced recurrence of uveitis at least 2 separate times requiring systemic, intra- or peri-ocular injection of corticosteroid.
4. At the time of enrollment (Day 1), the study eye has <10 anterior chamber cells/HPF (high power field) and a vitreous haze ≤ grade 2.
5. Visual acuity of study eye ≥15 letters on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
6. Not planning to undergo elective ocular surgery during the study.
7. Able to understand and sign the Informed Consent Form (ICF).
8. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Key Exclusion Criteria:

Ocular Exclusion Criteria (for the study eye, unless indicated otherwise):

1. History of posterior uveitis only that is not accompanied by vitritis or macular edema.
2. History of iritis only associated with no vitreous cells, anterior chamber cells, or vitreous haze at Day 1.
3. Uveitis with infectious etiology.
4. Vitreous hemorrhage.
5. Intraocular inflammation associated with a condition other than noninfectious uveitis (eg, intraocular lymphoma).
6. Uveitis limited to the anterior segment, ie, anterior uveitis only.
7. Ocular malignancy in either eye, including choroidal melanoma.
8. Previous viral retinitis.
9. Toxoplasmosis scar or scar related to previous viral retinitis in the study eye.
10. Current viral diseases of the cornea and conjunctiva including epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, and varicella, mycobacterial infections of the eye, or fungal diseases of ocular structures.
11. Media opacity precluding evaluation of retina and vitreous.
12. Peripheral retinal detachment in area of insertion.
13. Diagnosis of any form of glaucoma or ocular hypertension at Screening, unless previously treated with an incisional surgery procedure that has resulted in stable intraocular pressure (IOP) in the normal range [10-21 millimeter of mercury (mmHg)].
14. IOP >21 mmHg or concurrent therapy at Screening with any IOP lowering pharmacologic agent.
15. Chronic hypotony (<6 mmHg).
16. Ocular surgery within 12 weeks prior to Day 1.
17. Capsulotomy within 30 days prior to Day 1.
18. Prior intravitreal treatment with Retisert®, ILUVIEN®, or YUTIQ® (0.18 mg) within 156 weeks prior to Day 1.
19. Prior intravitreal treatment with OZURDEX® or sub-choroidal injection with XIPERE™ within 24 weeks prior to Day 1.
20. Prior intravitreal treatment with Triesence® or TRIVARIS™ within 12 weeks prior to Day 1.
21. Peri-ocular or subtenon steroid treatment within 12 weeks prior to Day 1.

    All other Exclusion Criteria:
22. Allergy to fluocinolone acetonide or any component of Yutiq 0.05 mg.
23. Requirement for chronic systemic or inhaled corticosteroid therapy (>15mg prednisone daily) or chronic systemic immunosuppressive therapy.
24. History of certain skin cancers (specifically, basal cell carcinoma and squamous cell carcinoma), any malignancy receiving treatment, or in remission less than 5 years prior to Day 1.
25. Positive test for human immunodeficiency virus (HIV) or syphilis during Screening.
26. Mycobacterial uveitis or chorioretinal changes of either eye which, in the opinion of the Investigator, result from infectious mycobacterial uveitis.
27. Systemic infection within 30 days prior to Day 1.
28. Any severe acute or chronic medical or psychiatric condition that could increase the risk associated with study participation or could interfere with the interpretation of study results and, in the judgment of the Investigator, could make the subject inappropriate for study enrollment.
29. Any other systemic or ocular condition which, in the judgment of the Investigator, could make the subject inappropriate for study enrollment.
30. Treatment with an investigational drug or device within 30 days prior to Day 1.
31. Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in the protocol from at least 14 days prior to Day 1 until the 52-week Visit.
32. Unlikely to comply with the study protocol or who are likely to be lost to follow-up within 52 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- EyePoint Study Site, Waltham, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3 prospective, controlled study was conducted in subjects with chronic non-infectious uveitis affecting the posterior segment of the eye at 8 sites in the United States between 13 October 2021 and 12 April 2023.
Pre-assignment Details: This study consists of a screening period (up to 30 days) and treatment period (52 weeks). A total of 12 subjects were enrolled in the study.
Units Other Than Participants: Eyes
Groups:
- Fluocinolone Acetonide 0.05 mg: Subjects received a single dose of intravitreal fluocinolone acetonide 0.05 mg on Day 1.
- Sham Injection: Subjects received a single intravitreal sham injection on Day 1.
Period: Overall Study
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Started | 6; 12 Eyes | 6; 12 Eyes
Completed | 6; 12 Eyes | 0; 0 Eyes
Not Completed | 0; 0 Eyes | 6; 12 Eyes
Not completed — Sponsor decided to stop study enrollment and terminate the study | 0 | 6

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) analysis set included all subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (12.48) | 51.7 (19.23) | 52.0 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 1 | 3
  White | 3 | 5 | 8
  Missing | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 3 | 4 | 7
  Not Stated | 1 | 0 | 1
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Recurrence of Uveitis in the Study Eye at Week 24
Description: Recurrence was defined as:
  * An increase in the vitreous haze of ≥2 steps compared to baseline or any visit time point prior to the Week 24 visit; or
  * A deterioration in visual acuity of at least 15 letters BCVA compared to baseline or any visit time point prior to the Week 24 visit.
Time Frame: Week 24
Population: The ITT analysis set included all subjects who were randomized. Data was not collected for Sham injection group due to early termination of study.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 6 | 0
percentage of subjects | 0 [0 to 45.9] |

2. Secondary Outcome: Percentage of Subjects With Recurrence of Uveitis in the Study Eye at Week 52
Description: Recurrence was defined as:
  * An increase in the vitreous haze of ≥2 steps compared to baseline or any visit time point prior to the Week 24 visit (or the Week 52 visit); or
  * A deterioration in visual acuity of at least 15 letters BCVA compared to baseline or any visit time point prior to the Week 24 visit (or the Week 52 visit).
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 6 | 0
percentage of subjects | 0 [0 to 45.9] |

3. Secondary Outcome: Percentage of Subjects With Recurrence of Uveitis in the Fellow Eye at Weeks 24 and 52
Description: as for outcome 2
Time Frame: Weeks 24 and 52
Population: Data was not collected for this outcome measure due to early termination of study.
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye at Weeks 24 and 52
Description: The BCVA was measured according to the standard procedure originally developed for Early Treatment Diabetic Retinopathy Study (ETDRS). The ETDRS letter score calculated when 20 or more letters were read correctly at 4.0 meters; the visual acuity letter score was equal to the total number of letters read correctly at 4.0 meters plus 30. The score ranges from 0 (worse) to 100 (best). Higher scores indicate positive outcome measure.
Time Frame: Weeks 24 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 6 | 0
score on a scale
  Week 24 | 9.7 (4.93) |
  Weeks 52 | 16.8 (12.11) |

5. Secondary Outcome: Number of Recurrences of Uveitis Within 24 and 52 Weeks
Description: Recurrence was defined as:
  An increase in the vitreous haze of ≥2 steps compared to baseline or any visit time point prior to the Week 24 visit (or the Week 52 visit); or A deterioration in visual acuity of at least 15 letters BCVA compared to baseline or any visit time point prior to the Week 24 visit (or the Week 52 visit).
Time Frame: Weeks 24 and 52
Population: as for outcome 1
Measure: Number; unit: recurrences of uveitis
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 6 | 0
recurrences of uveitis
  Week 24 | 0 |
  Week 52 | 0 |

6. Secondary Outcome: Time to Recurrence of Uveitis Through Weeks 24 and 52
Description: as for outcome 5
Time Frame: Weeks 24 and 52
Population: The ITT analysis set included all subjects who were randomized. Only subjects with recurrence of uveitis are reported. Data was not collected for Sham injection group due to early termination of study.
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Adjunctive Treatments Required to Treat Recurrences of Uveitis at 24 and 52 Weeks
Description: Recurrence was defined as:
  An increase in the vitreous haze of ≥2 steps compared to baseline or any visit time point prior to the Week 24 visit (or the Week 52 visit); or A deterioration in visual acuity of at least 15 letters BCVA compared to baseline or any visit time point prior to the Week 24 visit (or the Week 52 visit).
  In the event of a uveitis recurrence in either eye, peri-ocular or intraocular corticosteroid injections, or topical medications administered as first line local therapy.
Time Frame: Weeks 24 and 52
Population: as for outcome 6
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Subjects With Recurrence of Iridocyclitis in the Study Eye Compared to Baseline at 24 and 52 Weeks
Description: Iridocyclitis was defined as a >2-step increase in anterior chamber cells per high-power field (HPF) (1.6*using a 1-millimeter beam).
Time Frame: Weeks 24 and 52
Population: Data was not collected for this outcome measure due to early termination of study.
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Subjects With Resolution of Macular Edema at Day 28 and Months 2, 3, 6 and 12
Description: The macular edema was measured by spectral-domain - optical coherence tomography (SD-OCT) imaging.
Time Frame: At Day 28 and Months 2, 3, 6 and 12
Population: The ITT analysis set included all subjects who were randomized. Only subjects analyzed at specific timepoints are reported.
Measure: Number; unit: percentage of subjects
Arm/Group | Fluocinolone Acetonide 0.05 mg | Sham Injection
Number analyzed (Participants) | 6 | 6
percentage of subjects
  Day 28 - Yes: number analyzed (Participants) | 6 | 5
  Day 28 - Yes | 50.0 | 60.0
  Day 28 - No: number analyzed (Participants) | 6 | 5
  Day 28 - No | 50.0 | 40.0
  Month 2 - Yes: number analyzed (Participants) | 6 | 4
  Month 2 - Yes | 50.0 | 75.0
  Month 2 - No: number analyzed (Participants) | 6 | 4
  Month 2 - No | 50.0 | 25.0
  Month 3 - Yes: number analyzed (Participants) | 5 | 3
  Month 3 - Yes | 40.0 | 33.3
  Month 3 - No: number analyzed (Participants) | 5 | 3
  Month 3 - No | 60.0 | 66.7
  Month 6 - Yes: number analyzed (Participants) | 5 | 0
  Month 6 - Yes | 20.0 |
  Month 6 - No: number analyzed (Participants) | 5 | 0
  Month 6 - No | 80.0 |
  Month 12 - Yes: number analyzed (Participants) | 4 | 0
  Month 12 - Yes | 75.0 |
  Month 12 - No: number analyzed (Participants) | 4 | 0
  Month 12 - No | 25.0 |

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the study drug administration (Day 1) up to early termination of the study, approximately 52 weeks.
Description: The Safety Analysis Set included all subjects who were randomized and received fluocinolone acetonide 0.05 mg or sham injection.
Groups:
- Fluocinolone Acetonide 0.05 mg - Study Eye; Fluocinolone Acetonide 0.05 mg - Systemic: Subjects received a single dose of intravitreal fluocinolone acetonide 0.05 mg in study eye on Day 1.
- Fluocinolone Acetonide 0.05 mg - Fellow Eye: No study treatment administered in fellow eye.
- Sham Injection- Study Eye; Sham Injection- Systemic: Subjects received a single intravitreal sham injection in study eye on Day 1.
- Sham Injection- Fellow Eye: No sham treatment administered in fellow eye.
Arm/Group | Fluocinolone Acetonide 0.05 mg - Study Eye | Fluocinolone Acetonide 0.05 mg - Fellow Eye | Fluocinolone Acetonide 0.05 mg - Systemic | Sham Injection- Study Eye | Sham Injection- Fellow Eye | Sham Injection- Systemic
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 1/6 | 2/6 | 1/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide 0.05 mg - Study Eye (N=6) | Fluocinolone Acetonide 0.05 mg - Fellow Eye (N=6) | Fluocinolone Acetonide 0.05 mg - Systemic (N=6) | Sham Injection- Study Eye (N=6) | Sham Injection- Fellow Eye (N=6) | Sham Injection- Systemic (N=6)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluocinolone Acetonide 0.05 mg - Study Eye (N=6) | Fluocinolone Acetonide 0.05 mg - Fellow Eye (N=6) | Fluocinolone Acetonide 0.05 mg - Systemic (N=6) | Sham Injection- Study Eye (N=6) | Sham Injection- Fellow Eye (N=6) | Sham Injection- Systemic (N=6)
Epiretinal membrane (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Optic atrophy (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Posterior capsule opacification (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 0
Vitreal cells (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vitreous haze (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 1 | 0 | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Anterior chamber cell (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotony of eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The Sponsor made the decision to stop study enrollment and terminate the study for reasons other than safety or efficacy in early May 2022 upon receipt of FDA comments on the clinical program in January 2022.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT05070728/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT05070728/SAP_001.pdf